CLINICAL TRIAL: NCT06451510
Title: Knee Osteoarthritis in the Region of Norrbotten (KORN)
Brief Title: Knee Osteoarthritis in the Region of Norrbotten
Acronym: KORN
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Norrbotten (Unknown)
Responsible Party: Sponsor
Other Study IDs: DNR: 2016/20-31; SAR (Registry Identifier: Swedish Arthroplasty Register); SFR (Registry Identifier: Swedish Fracture Register)
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis; Knee Injuries; Knee Osteoarthritis; Tibial Plateau Fractures; Tibial Fractures; Patient Satisfaction; Quality of Life; Complication of Treatment
Keywords: Osteoarthritis; Knee; Tibial plateau fracture; Outcome; Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Knee Injuries; Osteoarthritis, Knee; Tibial Plateau Fractures; Tibial Fractures; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the prevalence of radiographic knee osteoarthritis and to report medium and long term functional outcomes secondary to tibia plateau fractures. The second aim was to investigate whether there were any risk factors associated with these outcomes.

DETAILED DESCRIPTION:
1. The study population consists of patients from the Swedish region of Norrbotten (northern part of Sweden) who had undergone TPF between the years of 2001 and 2015.
2. All patients are evaluated radiographically.
3. Condition-specific scores are assessed using the Knee injury and Osteoarthritis Outcome Score (KOOS). General health related quality of life are assessed by the EuroQol 5-Dimension 5-level (EQ-5D-5L) tool.
4. All patients are examined clinically.
5. The relationship between the development of radiographic OA in patients who had undergone TPF and such potential factors as gender, age, body mass index (BMI), fracture pattern or method of fracture treatment is being assessed.
6. The data from the Swedish Fracture Register and the Swedish Arthroplasty Register are used in order to follow the long-term results.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the region of Norrbotten (northern part of Sweden) who underwent tibial plateau fracture between the years of 2001 and 2015

Exclusion Criteria:

* Death without bilateral weighted X-ray minimum 5 years post injury
* Open growth plate in distal femur and/or proximal tibia
* Extraarticular or isolated eminentia fracture
* OA prior to injury
* Having a rheumatic disorder involving joints
* Earlier and/or later severe injury to the index knee
* Having cognitive disorders disqualifying from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consists the subjects who underwent tibial plateau fracture and that could be identified by a computer-assisted search of the local medical journal database Vård Administrativt System (VAS), using the ICD-10 diagnostic codes for proximal tibia fracture (open and closed) (S82.1, S82.8 and S 82.9).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with radiographic osteoarthritis (OA) | At least 5 years
  Number of participants with radiographic OA at follow-up at least five years after the tibial plateau fracture was considered the primary endpoint of this study.

SECONDARY OUTCOMES:
Score values in the condition-specific measure for assessment of symptoms and function related to the knee joint | At least 5 years
  The Knee injury and Osteoarthrtis Outcome Scale (KOOS) is used. KOOS is a self-administered knee-specific questionnaire consisting of 42 items in five subscales. A normalized score from 0 (extreme problems) to 100 (no problems at all) are calculated separately for each of the five subscales.
  Knee-related symptoms and function are evaluated with use of four out of five KOOS subscales: Pain, other Symptoms, Function in daily living (ADL) and Function in sport and recreation (Sport/Rec).
Score values in assessment of condition-specific health-related quality of life | At least 5 years
  The condition-specific measure, Knee injury and Osteoarthrtis Outcome Scale (KOOS) is used. The score values in the KOOS subscale knee-related Quality of Life (QOL) are evaluated.
Score values in assessment of general health-related qualilty of life | At least 5 years
  Assessment is performed with the EuroQol 5-Dimension 5-level (EQ-5D-5L). The questionnaire consists of five questions exploring five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels, ranging from "no problems" to "extreme problems". An EQ-5D-5L index of 1.0 indicates the best possible health state and 0.0 denotes death.

OTHER OUTCOMES:
Number of participants who had a surgical intervention due to OA secondary to the tibial plateau fracture | At least 5 years
  Number of participants who developed an end-stage OA and underwent either knee arthroplasty (either partial or total) or knee osteotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunderby Central Hospital of Norrbotten, Luleå, Norrbotten County, Sweden

REFERENCES:
- [Derived] Klaser J, Kotake L, Lindberg M, Wigge S, Lundqvist R, Szczesny G, Paradowski PT. Prevalence of osteoarthritis and clinical outcomes in patients with fractures of the tibial plateau - medium- and long-term analysis. BMC Musculoskelet Disord. 2025 May 27;26(1):522. doi: 10.1186/s12891-025-08786-7. PMID 40426131